CLINICAL TRIAL: NCT05349981
Title: Lyric Self-replacement Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: AccuData Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0700
Record Dates: First submitted 2021-09-28; First posted 2022-04-27 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Self-controlled repeated measures study design with a single cohort, intended to mimic clinical use case.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lyric self-replacement (Experimental): This cohort of experienced Lyric patients are required to meet the candidacy criteria to be eligible for the self-replacement procedure. They will also be required to demonstrate proficiency with the self-replacement procedure before proceeding with independent self-replacement.
  Interventions: Device: Phonak Lyric self-replacement procedure

INTERVENTIONS:
Device: Phonak Lyric self-replacement procedure — The self-replacement procedure is an experimental procedure in which the Lyric user replaces the Lyric devices independently at every other device replacement, using dedicated candidacy, training, and management procedures, conducted by and at the discretion of his/her hearing care provider (HCP).

SUMMARY:
This study is designed to investigate the effectiveness and safety of the Phonak Lyric self-replacement procedure, as compared to the HCP-replacement procedure.

ELIGIBILITY:
Inclusion Criteria:

* Meets requirements outlined on Lyric self-replacement candidacy form
* Current Lyric hearing instrument user with 3+ months of Lyric experience
* 22 years of age or older at the time of enrollment in the study
* Mild-to-moderately severe sensorineural hearing loss (bilaterally or unilaterally)
* Good understanding (read/write/speak) of the English language
* Willingness to comply with all study requirements

Exclusion Criteria:

* Does not meet requirements outlined on Lyric self-replacement candidacy form
* Difficulty understanding/reading instructions when corrected for vision loss
* Impairments that would restrict participation in any of the evaluations
* Ear health conditions present at baseline that prevent immediate device replacement
* Conditions that would indicate the need for medical referral prior to hearing aid fitting according to local regulations

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Change in aided audiometric threshold testing between standard and experimental replacement procedures | Baseline, during intervention, immediately after intervention
  Aided audiometric test measures: threshold testing. Thresholds will be measured in decibels Hearing Level (dBHL), with a range of -10 - 120 dBHL. Lower scores indicate better performance. Change in scores will be assessed between standard and experimental replacement procedures.
Change in aided speech-in-noise testing between standard and experimental replacement procedures | Baseline, during intervention, immediately after intervention
  Aided audiometric test measures: speech-in-noise testing. Scores will be measured using signal-to-noise ratio loss, with scores ranging from 0 - 25.5. Lower scores indicate better performance. Change in scores will be assessed between standard and experimental replacement procedures.

SECONDARY OUTCOMES:
Change in incidence of medical referrals secondary to device replacement procedure-related ear health outcome between standard and experimental replacement procedures | Through study completion, an average of 5 months
  Evaluation of incidence of medical referral secondary to device replacement, as determined necessary by the hearing care professional, and compared between the standard and experimental device replacement procedures

OTHER OUTCOMES:
Change in incidence of provider/clinical support needed across device replacement procedures | Through study completion, an average of 5 months
  Evaluation of incidence of provider/clinical support needed between device replacements, as recorded by study staff, and compared between time periods associated with the standard and experimental device replacement procedures
Change in incidence of acoustic feedback across device replacement procedures | Baseline, during intervention, immediately after intervention
  Evaluation of incidence of acoustic feedback secondary to device replacement, as subjectively reported by the end user, and compared between the standard and experimental device replacement procedures
Change in measured device position at replacement between standard and experimental replacement procedures | Baseline, during intervention, immediately after intervention
  Achieved insertion depth of device, as measured by the hearing care professional using the dedicated fitting tool, and compared between the standard and experimental fitting procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Gardner, AuD, Study Director — Sonova USA Inc
Locations (8):
- United States (8):
  - San Francisco Audiology, San Francisco, California
  - NYC Hearing Associates, New York, New York
  - Aim Hearing and Audiology, Greensboro, North Carolina
  - ENT & Audiology Associates, Raleigh, North Carolina
  - The Woodlands Hearing Center, The Woodlands, Texas
  - Bay Area Audiology and Hearing Aids, Webster, Texas
  - Richmond Hearing Doctors, Midlothian, Virginia
  - Richmond Hearing Doctors, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No